CLINICAL TRIAL: NCT01312961
Title: Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy, Safety, and Tolerability of SAR231893/REGN668 Administered Subcutaneously Once Weekly for 12 Weeks in Patients With Persistent Moderate to Severe Eosinophilic Asthma Who Are Partially Controlled/Uncontrolled by Inhaled Corticosteroid Plus Long-acting beta2 Agonist Therapy
Brief Title: Efficacy, Safety, and Tolerability of Dupilumab in Patients With Persistent Moderate to Severe Eosinophilic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT11457; U1111-1117-7826 (Other: UTN)
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab; Fluticasone; Albuterol; Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (for Dupilumab) (Placebo Comparator): Placebo (for Dupilumab) subcutaneous (SC) injection once weekly (qw) for 12 weeks added to background therapy of inhaled corticosteroids/long-acting beta2-adrenergic agonist (ICS/LABA) (Fluticasone/Salmeterol combination therapy at stable dose for 4 weeks followed by Fluticasone monotherapy, dose progressively decreased and discontinued at Week 9). Albuterol or Levalbuterol was given as rescue medication.
  Interventions: Drug: Placebo (for Dupilumab); Drug: Fluticasone/Salmeterol combination therapy; Drug: Fluticasone monotherapy; Drug: Albuterol; Drug: Levalbuterol
- Dupilumab 300 mg qw (Experimental): Dupilumab 300 mg SC injection qw for 12 weeks added to background therapy of ICS/LABA (Fluticasone/Salmeterol combination therapy at stable dose for 4 weeks followed by Fluticasone monotherapy, dose progressively decreased and discontinued at Week 9). Albuterol or Levalbuterol was given as rescue medication.
  Interventions: Drug: Dupilumab; Drug: Fluticasone/Salmeterol combination therapy; Drug: Fluticasone monotherapy; Drug: Albuterol; Drug: Levalbuterol

INTERVENTIONS:
Drug: Dupilumab — Solution for injection, one subcutaneous injection.
  Other Names: SAR231893; REGN668
  Arms: Dupilumab 300 mg qw
Drug: Placebo (for Dupilumab) — Solution for injection, one subcutaneous injection.
  Arms: Placebo (for Dupilumab)
Drug: Fluticasone/Salmeterol combination therapy — Oral inhalation twice daily.
Drug: Fluticasone monotherapy — Oral inhalation twice daily.
Drug: Albuterol — Oral inhalation as needed.
Drug: Levalbuterol — Oral inhalation as needed.

SUMMARY:
Primary Objective:

To investigate the effects of Dupilumab (SAR231893/REGN668) administered subcutaneously (SC) once weekly (qw) for 12 weeks as compared to placebo on reducing the incidence of asthma exacerbation in participants with persistent moderate to severe eosinophilic asthma.

Secondary Objectives:

* To assess the safety and tolerability of Dupilumab administered SC qw for 12 weeks in participants with persistent moderate to severe eosinophilic asthma.
* To assess Dupilumab serum concentrations following qw SC dosing for 12 weeks in participants with persistent moderate to severe eosinophilic asthma.

DETAILED DESCRIPTION:
The total duration of the study period per participant was 20-22 weeks broken down as follows:

* Screening period: up to 14 days,
* Treatment period: 12 weeks,
* Follow-up period: 6-8 weeks.

ELIGIBILITY:
Inclusion criteria:

Medical diagnosis of persistent asthma for at least 12 months whose:

* airway inflammation likely to be eosinophilic,
* asthma partially controlled or uncontrolled on ICS plus LABA therapy.
* On a stable dose of either Fluticasone/Salmeterol, Budesonide/Formoterol, Mometasone/Formoterol combination therapy for at least 1 month prior to screening.
* Signed an Informed Consent Form and Health Insurance Portability and Accountability Act (HIPAA) Authorization Form.

Exclusion criteria:

* Less than 18 years or greater than 65 years of age.
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further evaluation.
* Chronic obstructive pulmonary disease and/or other lung diseases impairing Pulmonary Function Tests.
* Beta-adrenergic receptor blockers required for any reason.
* Current smoker or cessation of smoking within the 6 months prior to screening.
* Previous smoking with a smoking history >10 cigarette pack/years.
* Participation in another study within 6 months prior to screening if the study medication was an antibody or within 30 days prior to screening for all other study medications.
* Known or suspected non-compliance, alcohol or drug abuse.
* Inability to follow the procedures of the study (e.g, due to language problems, psychological disorders).
* Concomitant severe diseases or diseases for which the use of ICS or LABA were contraindicated.
* Known allergy to doxycycline or related compounds.
* Pregnancy or intention to become pregnant during the course of the study, breast feeding, or unwillingness to use a highly effective method of contraception throughout the study in women of childbearing potential.
* Recent history of a parasitic infection or travel to a parasitic endemic area within 6 months prior to screening.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (50):
- United States (50):
  - Investigational Site Number 840047, Anaheim, California
  - Investigational Site Number 840046, Long Beach, California
  - Investigational Site Number 840032, Los Angeles, California
  - Investigational Site Number 840036, Los Angeles, California
  - Investigational Site Number 840005, Mission Viejo, California
  - Investigational Site Number 840007, Orange, California
  - Investigational Site Number 840048, Riverside, California
  - Investigational Site Number 840035, Rolling Hills Estates, California
  - Investigational Site Number 840041, San Francisco, California
  - Investigational Site Number 840042, San Francisco, California
  - Investigational Site Number 840039, San Jose, California
  - Investigational Site Number 840024, Santa Rosa, California
  - Investigational Site Number 840002, Stockton, California
  - Investigational Site Number 840031, Colorado Springs, Colorado
  - Investigational Site Number 840011, Denver, Colorado
  - Investigational Site Number 840017, Denver, Colorado
  - Investigational Site Number 840026, New Haven, Connecticut
  - Investigational Site Number 840044, Tallahassee, Florida
  - Investigational Site Number 840029, Tampa, Florida
  - Investigational Site Number 840028, Indianapolis, Indiana
  - Investigational Site Number 840038, Iowa City, Iowa
  - Investigational Site Number 840021, Overland Park, Kansas
  - Investigational Site Number 840053, Owensboro, Kentucky
  - Investigational Site Number 840014, Baltimore, Maryland
  - Investigational Site Number 840015, North Dartmouth, Massachusetts
  - Investigational Site Number 840003, Minneapolis, Minnesota
  - Investigational Site Number 840010, Minneapolis, Minnesota
  - Investigational Site Number 840006, St Louis, Missouri
  - Investigational Site Number 840013, St Louis, Missouri
  - Investigational Site Number 840022, Bozeman, Montana
  - Investigational Site Number 840025, Omaha, Nebraska
  - Investigational Site Number 840008, Papillion, Nebraska
  - Investigational Site Number 840018, Princeton, New Jersey
  - Investigational Site Number 840004, Winston-Salem, North Carolina
  - Investigational Site Number 840023, Sylvania, Ohio
  - Investigational Site Number 840045, Oklahoma City, Oklahoma
  - Investigational Site Number 840001, Lake Oswego, Oregon
  - Investigational Site Number 840012, Medford, Oregon
  - Investigational Site Number 840016, Portland, Oregon
  - Investigational Site Number 840040, Hershey, Pennsylvania
  - Investigational Site Number 840037, Pittsburgh, Pennsylvania
  - Investigational Site Number 840009, Upland, Pennsylvania
  - Investigational Site Number 840027, Charleston, South Carolina
  - Investigational Site Number 840030, El Paso, Texas
  - Investigational Site Number 840050, San Antonio, Texas
  - Investigational Site Number 840052, South Burlington, Vermont
  - Investigational Site Number 840049, Richmond, Virginia
  - Investigational Site Number 840020, Seattle, Washington
  - Investigational Site Number 840019, Tacoma, Washington
  - Investigational Site Number 840034, Madison, Wisconsin

REFERENCES:
- [Result] Wenzel S, Ford L, Pearlman D, Spector S, Sher L, Skobieranda F, Wang L, Kirkesseli S, Rocklin R, Bock B, Hamilton J, Ming JE, Radin A, Stahl N, Yancopoulos GD, Graham N, Pirozzi G. Dupilumab in persistent asthma with elevated eosinophil levels. N Engl J Med. 2013 Jun 27;368(26):2455-66. doi: 10.1056/NEJMoa1304048. Epub 2013 May 21. PMID 23688323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 50 sites in the United States. A total of 491 participants were screened between March 2011 and June 2012, of whom 104 were randomized at 28 sites. A total of 387 participants were screen failures mainly due to inclusion criteria for eosinophilic asthma not met.
Pre-assignment Details: Randomization was stratified according to prior inhaled corticosteroids/long-acting beta2-adrenergic agonist (ICS/LABA) combination therapy dose. Assignment to arms was done centrally using Interactive Voice Response System in 1:1 ratio to receive either Dupilumab 300 mg or Placebo.
Groups:
- Placebo (for Dupilumab): Placebo (for Dupilumab) subcutaneous (SC) injection once weekly (qw) for 12 weeks added to background therapy of ICS/LABA (Fluticasone/Salmeterol combination therapy at stable dose for 4 weeks followed by Fluticasone monotherapy, dose progressively decreased and discontinued at Week 9). Albuterol or Levalbuterol were given as rescue medication.
Period: Overall Study
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Started | 52 | 52
Treated | 52 | 52
Completed | 35 | 45
Not Completed | 17 | 7
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 11 | 1
Not completed — Poor compliance to protocol | 1 | 0
Not completed — Other than specified above | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline participants included all randomized participants.
Groups:
- Placebo (for Dupilumab): Placebo (for Dupilumab) SC injection qw for 12 weeks added to background therapy of ICS/LABA (Fluticasone/Salmeterol combination therapy at stable dose for 4 weeks followed by Fluticasone monotherapy, dose progressively decreased and discontinued at Week 9). Albuterol or Levalbuterol were given as rescue medication.
- Total: Total of all reporting groups
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (13.1) | 37.8 (13.2) | 39.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 26 | 26 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 12 | 16
  Not Hispanic or Latino | 48 | 40 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  Caucasian/White | 38 | 45 | 83
  Black | 9 | 5 | 14
  Asian/Oriental | 3 | 1 | 4
  Other than specified above | 2 | 1 | 3
Prior ICS/LABA Combination Therapy Dose [Count of Participants; unit: Participants] — High-Dose combination therapy was defined as Fluticasone (≥500 µg) and Salmeterol (50 µg) twice daily or the equivalent. Medium-dose combination therapy was defined as Fluticasone (250-499 µg) and Salmeterol (50 µg) twice daily or the equivalent.
  Participants
    High Dose | 41 | 42 | 83
    Medium Dose | 11 | 10 | 21
Morning Peak Expiratory Flow (PEF) [Mean (Standard Deviation); unit: L/min] — PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. Testing for PEF was performed at home while sitting or standing prior to using any medication for asthma. Population: Number of participants analyzed = participants with available data for this baseline measure.
  L/min
    number analyzed (Participants) | 52 | 51 | 103
    (all) | 406.87 (110.74) | 393.04 (101.13) | 400.02 (105.80)
Number of Inhalations of Albuterol or Levalbuterol in a 24-hour Period [Mean (Standard Deviation); unit: number of inhalations] — Number of Albuterol or Levalbuterol inhalations were recorded daily by the participants in their electronic diary. Population: Number of participants analyzed = participants with available data for this baseline measure.
  number of inhalations
    number analyzed (Participants) | 52 | 50 | 102
    (all) | 2.04 (1.78) | 2.16 (2.40) | 2.10 (2.10)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Asthma Exacerbation
Description: An asthma exacerbation was defined as the occurrence of any of the following: ≥30% reduction from baseline in morning PEF on 2 consecutive days; or ≥6 additional reliever puffs of albuterol or levalbuterol in a 24-hour period (compared to baseline) on 2 consecutive days; or deterioration of asthma, as determined by the investigator, requiring systemic steroid treatment, or an increase in inhaled corticosteroid (ICS) of ≥4 times the last dose received prior to discontinuation from the study, or hospitalization. The occurrence of asthma exacerbations by individual criteria are reported.
Time Frame: Baseline up to Week 12
Population: Modified intent-to-treat (mITT) population that included all randomized participants who received at least one dose of study drug. Participants were analysed in the treatment group to which they were randomized.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (for Dupilumab): Placebo (for Dupilumab) SC injection qw for 12 weeks added to background therapy of ICS/LABA (Fluticasone/Salmeterol combination therapy at stable dose for 4 weeks followed by Fluticasone monotherapy, dose progressively decreased and discontinued at Week 9). Albuterol or Levalbuterol was given as rescue medication.
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 52 | 52
percentage of participants
  Asthma exacerbation | 44.2 | 5.8
  ≥30% reduction from baseline in morning PEF | 19.2 | 1.9
  ≥6additional albuterol/levalbuterol puffs | 19.2 | 1.9
  Systemic steroid treatment | 9.6 | 1.9
  Increase in ICS ≥4 times baseline dose of ICS | 5.8 | 0.0
  Hospitalization | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo (for Dupilumab) vs Dupilumab 300 mg qw; Analysis was performed using a logistic regression model with treatment groups and stratification factor (prior ICS/LABA combination therapy dose) as covariates; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.077, 95% CI 2-sided [0.021 to 0.280] — Dupilumab 300 mg vs. Placebo

2. Secondary Outcome: Time to First Asthma Exacerbation: Kaplan-Meier Estimates at Week 4, Week 8 and Week 12
Description: The time-to-asthma exacerbation was defined as the time from the date of randomization to the date of the first asthma exacerbation event; for participants without asthma exacerbation, it was censored at the end of treatment visit date. The median time to first asthma exacerbation was not estimated because the number of asthma exacerbations was too low in the Dupilumab arm. Therefore, alternative Kaplan-Meier statistics, the probability of asthma exacerbation at Week 4, 8 and 12, are presented as the descriptive measure statistics.
Time Frame: Baseline up to Week 12
Population: mITT population.
Measure: Number (95% Confidence Interval); unit: Probability of asthma exacerbation
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 52 | 52
Probability of asthma exacerbation
  Probability at Week 4 | 0.058 [0.000 to 0.122] | 0.038 [0.000 to 0.091]
  Probability at Week 8 | 0.245 [0.124 to 0.366] | 0.058 [0.000 to 0.121]
  Probability at Week 12 | 0.460 [0.318 to 0.602] | 0.058 [0.000 to 0.121]

3. Secondary Outcome: Percentage of Participants With Composite Asthma Events
Description: Composite asthma event was defined as a 30% or greater reduction from baseline in morning PEF on 2 consecutive days together with 6 or more additional reliever puffs of albuterol or levalbuterol in a 24-hour period (compared to baseline) on 2 consecutive days.
Time Frame: Baseline up to Week 12
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 52 | 52
percentage of participants | 1.9 | 0

4. Secondary Outcome: Change From Baseline in Forced Expiratory Flow in One Second (FEV1) to Week 12
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: Baseline, Week 12
Population: mITT population. Number of participants analyzed = participants with at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Placebo: Placebo (for Dupilumab) SC injection qw for 12 weeks added to background therapy of ICS/LABA (Fluticasone/Salmeterol combination therapy at stable dose for 4 weeks followed by Fluticasone monotherapy, dose progressively decreased and discontinued at Week 9). Albuterol or Levalbuterol was given as rescue medication.
Arm/Group | Placebo | Dupilumab 300 mg qw
Number analyzed (Participants) | 36 | 45
Liters | -0.12 (0.35) | 0.06 (0.32)

5. Secondary Outcome: Change From Baseline in Peak Expiratory Flow (PEF) to Week 12
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. Peak flow testing for PEF was performed at home (morning and evening) while sitting or standing prior to using any medication (if needed) for asthma.
Time Frame: Baseline, Week 12
Population: mITT population. Number analyzed = participants with at least one post-baseline assessment for each category.
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 52 | 52
liters/minute
  Change in morning PEF: number analyzed (Participants) | 36 | 44
  Change in morning PEF | -11.2 (66.1) | 10.6 (48.5)
  Change in evening PEF: number analyzed (Participants) | 35 | 45
  Change in evening PEF | -15.6 (70.7) | -3.4 (49.3)

6. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (5-question Version [ACQ-5]) to Week 12
Description: ACQ-5 questionnaire is a validated questionnaire comprising of 5 questions for asthma symptoms: woken at night by symptoms, wake in the mornings with symptoms, limitation of daily activities, shortness of breath, and wheeze. Participants were asked to rate their asthma symptoms during the previous week on a 7-point scale as 0=no impairment, 6=maximum impairment. ACQ-5 score is the mean of the 5 questions and range between 0 (disease totally controlled) and 6 (disease severely uncontrolled), a higher score indicated lower asthma control.
Time Frame: Baseline, Week 12
Population: mITT population. Number of participants analyzed = participants with at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 36 | 44
units on a scale | -0.50 (1.12) | -1.07 (0.94)

7. Secondary Outcome: Change From Baseline in 22-item Sinonasal Outcome Test (SNOT-22) Score to Week 12
Description: The SNOT-22 is a validated measure of health related quality of life in sinonasal disease. It is a 22 item questionnaire with each item assigned a score ranging from 0-5. The total score may range from 0 (no disease) -110 (worst disease), lower scores represent better health related quality of life.
Time Frame: Baseline, Week 12
Population: mITT population. Number of participants analyzed = participants with at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 51 | 50
units on a scale | 1.27 (15.85) | -9.17 (15.40)

8. Secondary Outcome: Change From Baseline in Morning Asthma Symptom Scores to Week 12
Description: AM (ante meridiem) symptom scoring system rates were participant's overall asthma symptoms experienced during the night. It ranges from 0 to 4 as: 0 = No asthma symptoms, slept through the night, 1= Slept well, but some complaints in the morning. No nighttime awakenings,2= Woke up once because of asthma (including early awakening),3= Woke up several times because of asthma (including early awakening), 4= Bad night, awake most of the night because of asthma.
Time Frame: Baseline, Week 12
Population: mITT population. Number of participants analyzed = participants with at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 36 | 45
units on a scale | 0.3 (0.7) | -0.4 (0.7)

9. Secondary Outcome: Change From Baseline in Evening Asthma Symptom Scores to Week 12
Description: PM (post meridiem) symptom scoring system rates were participant's overall asthma symptoms experienced during the day. It ranges from 0 to 4 as: 0=very well, no asthma symptoms, 1=one episode of wheezing, cough, or breathlessness, 2=more than one episode of wheezing, cough, or breathlessness without interference of normal activities, 3=wheezing, cough, or breathlessness most of the day, which interfered to some extent with normal activities, 4=asthma very bad, unable to carry out daily activities as usual.
Time Frame: Baseline, Week 12
Population: mITT population. Number of participants analyzed = participants with at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 36 | 45
units on a scale | 0.1 (0.9) | -0.5 (0.6)

10. Secondary Outcome: Change From Baseline in Number of Nocturnal Awakenings Per Day to Week 12
Description: Participants recorded every morning on awakening the number of asthma-related nocturnal awakenings requiring use of rescue medication that occurred during the previous night.
Time Frame: Baseline, Week 12
Population: mITT population. Number of participants analyzed = participants with at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: number of awakenings/day
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 36 | 45
number of awakenings/day | 0.1 (0.7) | -0.3 (0.7)

11. Secondary Outcome: Change From Baseline in Number of Inhalations Per Day of Albuterol or Levalbuterol to Week 12
Description: Number of Albuterol or Levalbuterol inhalations were recorded daily by the participants in their electronic diary as Albuterol or Levalbuterol was to be used only as needed for symptoms, not on a regular basis or prophylactically.
Time Frame: Baseline, Week 12
Population: mITT population. Number of participants analyzed = participants with at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: number of inhalations/day
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
Number analyzed (Participants) | 36 | 44
number of inhalations/day | 0.4 (2.4) | -1.3 (1.7)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 20) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment emergent AEs that developed/worsened and deaths that occurred during the 'on treatment period' (time from first dose of investigatory medicinal product (IMP) up to the end of the follow-up period [i.e. up to 7 weeks after the last dose of IMP]).
Groups:
- Placebo (for Dupilumab): Participants exposed to Placebo (for Dupilumab) SC injection qw for 12 weeks added to background therapy of ICS/LABA (mean exposure of 11 weeks).
- Dupilumab 300 mg qw: Participants exposed to Dupilumab 300 mg SC injection qw for 12 weeks added to background therapy of ICS/LABA (mean exposure of 11 weeks).
Arm/Group | Placebo (for Dupilumab) | Dupilumab 300 mg qw
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 3/52 | 1/52
Other Adverse Events (participants affected / at risk) | 24/52 | 33/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (for Dupilumab) (N=52) | Dupilumab 300 mg qw (N=52)
Pneumonia (Infections and infestations) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (for Dupilumab) (N=52) | Dupilumab 300 mg qw (N=52)
Gastroenteritis viral (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 7
Sinusitis (Infections and infestations) | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 7
Viral upper respiratory tract infection (Infections and infestations) | 0 | 3
Headache (Nervous system disorders) | 3 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3
Injection site erythema (General disorders) | 0 | 3
Injection site pain (General disorders) | 3 | 5
Injection site rash (General disorders) | 0 | 3
Injection site reaction (General disorders) | 0 | 5
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.